CLINICAL TRIAL: NCT06803108
Title: Pyramidal Versus Continuous Training Effects on Fatty Liver
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of physical therapy for Cardiovascular, Respiratory disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.R.E.C/012/004669
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group number 1 (Experimental): this group of this study will be fatty liver subjects (19 subjects in this group). . In this group, a pyramidal training will be adopted for nearly 60 minutes (nearly two rounds of 21 minutes of running on electronic treadmill will be separated with 10 minutes of rest between the two rounds. Also, warming (4 minutes before start of pyrimidal trianing) and cooling (4 minutes after pyramidal training) will be done through gentle stretching exercises/activities. the form of exercise will be done three times per week. the total study time will be 12 weeks. to be mentioned , this group will follow low calorie diet
  Interventions: Behavioral: pyramidal activity program
- group number 2 (Experimental): this group of this study will be fatty liver subjects (19 subjects). aerobic training on electronic treadmill will be adopted for 60 minutes in this group with moderate intensity. this form of exercise will be done three times per week. the total study time will be 12 weeks. to be mentioned , this group will follow low clorie diet
  Interventions: Behavioral: aerobic activity program

INTERVENTIONS:
Behavioral: pyramidal activity program — the participating subjects of this group of this study will be fatty liver subjects (19 subjects in this group). aerobic training on electronic treadmill will be adopted for 60 minutes in one group. In this group, a pyramidal training will be adopted for nearly 60 minutes (nearly two rounds of 21 minutes of running on electronic treadmill will be separated with 10 minutes of rest between the two rounds. Also, warming (4 minutes before start of pyrimidal trianing) and cooling (4 minutes after pyramidal training) will be done through gentle stretching exercises/activities. this form form of exercise will be done three times per week. the total study time will be 12 weeks. to be mentioned, the this group will follow low clorie diet
  Arms: group number 1
Behavioral: aerobic activity program — the participating subjects of the this group of this study will be fatty liver subjects (19 subjects in this group). aerobic training on electronic treadmill will be adopted for 60 minutes in this group with moderate intensity. the form of exercise will be done three times per week. the total study time will be 12 weeks. to be mentioned , this group will follow low clorie diet
  Arms: group number 2

SUMMARY:
exercise is very important maneuver in the control of elevated liver enzymes in complaint of fatty liver .. the exercise forma are many.. from these exercises, pyramidal training or continues aerobic one.

DETAILED DESCRIPTION:
the total participating subjects of the two groups of this study will be fatty liver subjects (19 subjects in every group). aerobic training on electronic treadmill will be adopted for 60 minutes in one group. In the other group, a pyramidal training will be adopted for nearly 60 minutes (nearly two rounds of 21 minutes of running on electronic treadmill will be separated with 10 minutes of rest between the two rounds. Also, warming (4 minutes before start of pyrimidal trianing) and cooling (4 minutes after pyramidal training) will be done through gentle stretching exercises/activities. the both forms of exercises will be done three times per week. the total study time will be 12 weeks. to be mentioned , the two groups followed low clorie diet

ELIGIBILITY:
Inclusion Criteria:

* fatty liver patients
* obese patients
* all patients will class one obesity

Exclusion Criteria:

* cardiovascular complaint
* metabolic complaints
* othopedic pains in lower limbs

Ages: 37 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — self-representation of gender identity.
Enrollment: 38 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
alanine transamianse | it will be measured after 12 weeks
  it is a liver enzyme

SECONDARY OUTCOMES:
aspartate transaminase | it will be measured after 12 weeks
  it is a liver enzyme
alkaline phosphatase | it will be measured after 12 weeks
  it is a liver enzyme
Gamma-glutamyl transferase | it will be measured after 12 weeks
  it is a liver enzyme
triglycerides | it will be measured after 12 weeks
  it will measured in serum
high density lipoprotein | it will be measured after 12 weeks
  it will measured in serum
body mass index | It will be measured after 12 weeks
  it will be measured on empty stomach
waist circumference | It will be measured after 12 weeks
  it will be measured at level of umbilicus

CONTACTS AND LOCATIONS:
Overall Officials: Ali MA Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo Unoversity, Giza, Egypt